CLINICAL TRIAL: NCT03566407
Title: Blood and Stool Molecular Biomarkers Longitudinal Detection Study in Crohn's Disease (CD) Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor decided to discontinue the study due to poor enrollment.
Sponsor: Prometheus Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 17IBD01
Record Dates: First submitted 2018-04-02; First posted 2018-06-25 (Actual); Last update posted 2019-06-07 (Actual); Status verified 2019-06

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — Colonoscopy

STUDY DESIGN:
Intervention Model Description: All study subjects will undergo a protocol required 6 month colonoscopy
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Group (Other): This is a prospective, longitudinal descriptive study of subjects with diagnosed Crohn's disease. Blood samples for measurement of protein biomarkers (serology), fresh whole blood for detection of gene polymorphisms, and stool samples for detection and assessment of microbiome and host DNA will be collected, and colonoscopy will be performed.
  Interventions: Procedure: Colonoscopy

INTERVENTIONS:
Procedure: Colonoscopy — Colonoscopy will be required for all subjects at 6 months - Visit 3.

SUMMARY:
To evaluate the relationship between noninvasive biomarkers (patient serological markers and metagenomic analysis of stool) and disease status as determined by colonoscopy and by clinical symptoms in patients with Crohn's disease, and to evaluate whether changes in the biomarker levels over time correlate to changes in the state of patients' disease.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females with CD who are 18 years of age or older on the date of obtaining informed consent and are undergoing a colonoscopy at the study site.
2. The patient must have a confirmed diagnosis of CD based on results a complete medical evaluation and the assessment by a physician specialized in inflammatory bowel disease.
3. All CD patients should have no evidence for another active organic disease of the GI tract or medical problems as specified below in the exclusion criteria.
4. All patients must have a colonoscopic examination performed preferably on the same day as blood specimen is drawn, or blood may be drawn up to one week prior to colonoscopy. Stool specimen will be collected prior to the beginning of bowel prep for the colonoscopy, up to 10 days prior to bowel prep.
5. Understand the procedures and requirements of the study by providing written informed consent including consent and authorization for protected health information disclosure.

Exclusion Criteria:

1. Extensive small bowel resection or short bowel syndrome.
2. Surgery for CD within the 6 months previous to enrollment.
3. Receipt of any blood products within 3 months prior to study entry.
4. Known pregnancy or breast feeding within 3 months of specimen collection.
5. Recent history of viral or bacterial gastroenteritis including Clostridium difficile infection < 4 weeks prior to the blood draw
6. Concurrent diagnosis of another currently active erosive GI mucosal disease such as erosive esophagitis, gastric or duodenal ulcer, celiac sprue, diverticulitis, etc.
7. History of intestinal or colorectal cancer, of active autoimmune diseases, or of other chronic uncontrolled systemic disorders
8. History of bowel prep within the past 3 months.
9. History of alcohol or substance abuse.
10. History of prior colectomy or stricturing disease that could limit colonoscopy examination of small bowel mucosa.
11. Current ostomy or ileoanal pouch.
12. Current or previous (of less than 4 weeks prior) participation in in a clinical trial for an investigational drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2018-05-04 (Actual); Primary Completion 2019-03-29 (Actual); Study Completion 2019-03-29 (Actual)

PRIMARY OUTCOMES:
Assess disease status biomarkers against colonoscopy | 6 months
  The primary endpoint for assessing clinical validity of candidate biomarker will be correlation to the degree of mucosal healing as determined by colonoscopy scored by the Simple Endoscopic Score for Crohn's Disease (SES-CD). - A scale that via colonoscopy of Crohn's disease patients measures: 1. Presence and size of ulcers 2. Extent of ulcerated surface 3. Extent of affected surface and 4. Presence and type of intestinal narrowings. Scale goes from 0 to 56 with a higher score indicating greater severity of disease.
Assess disease status biomarkers against colonoscopy | 6 months
  The primary endpoint for assessing clinical validity of candidate biomarker will also be correlated to the degree of mucosal healing as determined by colonoscopy scored by the Crohn's Disease Endoscopic Index of Severity (CDEIS). A scale that via colonoscopy of Crohn's disease patient's measures: 1. Deep Ulcerations 2. Superficial Ulcerations 3. Surface involved by disease and 4.Surface involved by ulcerations. Scale goes from 0 to 44 with a higher score indicating greater severity of disease.

SECONDARY OUTCOMES:
Assess bacterial markers in stool against colonoscopy scoring system Simple Endoscopic Score for Crohn's Disease (SES-CD) | 6 months
  Identify the correlation of the quantity of specific bacterial markers in the stool as quantified by a stool-based algorithm to the clinical state of the colonoscopy procedure scored by SES-CD tool. Simple Endoscopic Score for Crohn's Disease (SES-CD) - A scale that via colonoscopy of Crohn's disease patients measures: 1.Presence and size of ulcers 2. Extent of ulcerated surface 3. Extent of affected surface and 4. Presence and type of intestinal narrowings. Scale goes from 0 to 56 with a higher score indicating greater severity of disease.
Assess bacterial markers in stool against colonoscopy scoring system Crohn's Disease Endoscopic Index of Severity (CDEIS) | 6 months
  Identify the correlation of the quantity of specific bacterial markers in the stool as quantified by a stool-based algorithm to the clinical state of the colonoscopy procedure scored by CDEIS tool. Crohn's Disease Endoscopic Index of Severity (CDEIS) ) - A scale that via colonoscopy of Crohn's disease patient's measures: 1. Deep Ulcerations 2. Superficial Ulcerations 3. Surface involved by disease and 4.Surface involved by ulcerations. Scale goes from 0 to 44 with a higher score indicating greater severity of disease.
Assess bacterial markers in stool against disease symptomology scored by Harvey Bradshaw Index (HBI) for clinical evaluation | 6 months
  Determine the correlation of the quantity of specific bacterial markers in the stool as quantified by a stool-based algorithm to the clinical symptoms that measure stool frequency and symptomology by the Harvey Bradshaw Index (HBI) tool. Harvey Bradshaw Index (HBI) - A scale that assesses Crohn's disease patients' signs and symptoms by measuring : 1. General well-being 2. Abdominal pain 3. Number of liquid stools per day 4. Presence of abdominal mass and 5. Complications. Scale goes from 0 to 18 with a higher score indicating greater severity of disease.
Assess bacterial markers in stool against disease symptomology scored by Crohn's Disease Activity Index (CDAI) for clinical evaluation | 6 months
  Determine the correlation of the quantity of specific bacterial markers in the stool as quantified by a stool-based algorithm to the clinical symptoms that measure stool frequency and symptomology by the Crohn's Disease Activity Index (CDAI) tool. Crohn's Disease Activity Index (CDAI) - A scale that assesses Crohn's disease patients' signs and symptoms by measuring: 1. Number of liquid or soft stools each day for seven days 2. Abdominal pain each day for seven day 3. General well-being, subjectively assessed for day for seven days 4. Presence of complications 5. Taking anti-diarrhea medications 6. Presence of an abdominal mass 7.Hematocrit and 8. Percentage deviation from standard weight. Scale goes from 0 to >600 with a higher score indicating greater severity of disease.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development and Medical Affairs, Study Chair — Prometheus Laboratories
Locations (5):
- United States (5):
  - University of Southern California, Los Angeles, California
  - Ventura Clinical Trials, LLC., Ventura, California
  - Medical Research Center of Connecticut, LLC, Hamden, Connecticut
  - Atlanta Gastroenterology Associates, LLC, Atlanta, Georgia
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided